CLINICAL TRIAL: NCT06702163
Title: The Effects of EXOPULSE Mollii Suit on Motor Functions in Patients with Stroke (EXOSTROKE)
Brief Title: EXOPULSE Mollii Suit, Motor Function & Stroke (EXOSTROKE)
Acronym: EXOSTROKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut De La Colonne Vertebrale Et Des Neurosciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-A00232-41
Record Dates: First submitted 2024-11-03; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-02

CONDITIONS: Spasticity As Sequela of Stroke
Keywords: EXOPULSE Mollii Suit; Motor Functions & Stroke; Spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: We designed a randomized crossover, sham-controlled, double blind trial to demonstrate the improvement of motor functions and stroke related symptoms following a single session of "active" versus "sham" EXOPULSE Mollii suit. A 2-week washout period should be enough to prevent a potential carry over effect.
  Two weeks after the end of this phase (phase 1), a second phase of this trial, an open label phase, will be proposed for all patients to understand the effects of EXOPULSE Mollii suit employed over 4 weeks (a session every other day for a total of 14 sessions) on stroke related symptoms.
  Summary:
  * Phase 1: randomized sham-controlled crossover study (active versus sham condition)
  * Phase 2: Open-label study (active condition)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Condition (Active Comparator): Active sessions will last 1 hour each. The following parameters will be used for electric stimulation: low frequency (20 Hz), low current intensity (2 mA), with a small pulse width of 25-170 microseconds. These parameters were previously found to be safe in human studies. Based on the clinical exam of each patient, the spastic muscles will be targeted.
  EXOPULSE Mollii Suit is used for activation of weak muscles or relaxation of spastic muscles mediated by a physiological reflex mechanism referred to as reciprocal inhibition. By sending an electrical signal to an antagonistic muscle, the spastic muscle will subsequently relax.
  Interventions: Device: EXOPULSE MOLLII SUIT (active)
- Control Condition (Sham Comparator): In the control condition, the patients will receive a sham stimulation, for which the control unit will be programmed to start stimulating for 1 minute then it will shut off. There is no risk related to the sham intervention since it consists of applying the same parameters used for the active session (low frequency: 20 Hz; current intensity: 2 mA; pulse width ranging from 25 to 170 µs) but for a shorter duration of time (1 minute instead of 1 hour).
  Interventions: Device: EXOPULSE MOLLII SUIT (sham)

INTERVENTIONS:
Device: EXOPULSE MOLLII SUIT (active) — Exopulse Mollii suit is a new assistive device that has been developed by Exoneural Network (initially Inerventions AB), a Swedish med-tech company.
  Exopulse Mollii suit is a full-body garment with integrated 58 electrodes that can transcutaneously stimulate several groups of muscles. This stimulation is not intended to obtain a motor effect (contraction of the muscles in question), but rather to decrease the spasticity in spastic muscles by activating the antagonistic muscles via the physiological mechanism of reciprocal inhibition. The device is CE labelled and is intended to use for reducing spasticity and improving blood circulation. The outfit is very easy to put on, it can be used for one hour every day and the analgesic effects last 24 hours or more.
  Arms: Experimental Condition
Device: EXOPULSE MOLLII SUIT (sham) — In the sham condition, the control unit will be programmed to start stimulating for 1 minute then it will shut off.
  Arms: Control Condition

SUMMARY:
Spasticity is a common and debilitating complication in neurological conditions such as multiple sclerosis, cerebral palsy, and stroke. Stroke, a leading cause of global disability and death, occurs when blood flow to the brain is disrupted, causing neuronal damage. Approximately 80% of strokes are ischemic, with 20% being hemorrhagic. Several factors, including age, sex, vascular conditions, and lifestyle choices, increase the risk of stroke. Spasticity affects 19-28% of stroke survivors in the short term and up to 46% in the long term, severely impacting mobility and quality of life. Management typically involves pharmacological and nonpharmacological interventions, though these often have limited effectiveness and side effects. In this context, non-invasive techniques like transcutaneous stimulation with the EXOPULSE Mollii suit may offer a valuable alternative for managing spasticity and its associated symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years.
* Having a clinical diagnosis of stroke for at least three months
* Being able to walk freely or with the need of support (modified Rankin score

  * 4)
* Being a French speaker, able to understand verbal instructions, and affiliated with the national health insurance (sécurité social).
* Having spasticity with a score of at least 1+ on the MAS

Exclusion Criteria:

* Being included in another research protocol during the study period.
* Inability to undergo medical monitor for the study purposes due to geographical or social reasons.
* Having contraindications for using EXOPULSE Mollii suit (having implanted electronic medical devices or equipment which can be disrupted by magnets or an electronic life support equipment or high-frequency operation equipment; e.g., cardiac stimulator, ventriculoperitoneal shunt, intrathecal baclofen pump).
* Being pregnant (confirmed by a blood beta-HCG test).
* Having a change in their pharmacological therapy in the last three months.
* Suffering from other somatic or neuropsychiatric diagnoses (e.g., arrhythmias, uncontrolled epilepsy, diseases causing osteoarticular and muscular pain).
* Having a body mass index above 35 Kg/m2.
* In case of introducing a medical device other than EXOPULSE Mollii suit during the study period.
* Patients under juridical protection (" mesure de protection) judiciare : tutelle, curatelle, sauvegarde de justice ")
* Patients deprived of freedom (" personnes privées de liberté ".)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in balance using the BBS (Berg Balance Scale) ) before and after active and sham stimulation | This will be assessed before and after each condition (phase 1, 1 session per condition sham or active stimulation) on Day 0 (Visit1), Day 15 (Visit2), Day 30 (Visit3) and Day 45 (Visit4)
  Balance will be assessed using the 14-item BBS which has good psychometric properties in patients with stroke. The scale rates the balance using 56 points, with higher scores indicating better balance abilities. A score equal to or below 45 is commonly associated with the risk of falls across the literature.

SECONDARY OUTCOMES:
Assessment of the cumulative effects of EXOPULSE Mollii suit on balance using the BBS (Berg Balance Scale) | Evaluation will occur before Visit 5 (Day 60) and after Visit 6 (Day 90) 4 weeks of using EXOPULSE Mollii suit
  The cumulative effects of EXOPULSE Mollii Suit will be assessed following 4 weeks of using the device (3-4 times per week, during the open-label phase 2)
Assessment of the spasticity using the MAS (Modified Ashworth Scale) and the VAS pain (Visual Analogue Scale) | This will be assessed through study completion, an average of 3 months (at Visits 1, 2, 3, 4, 5 and 6)
  Spasticity will be evaluated by examiners using the MAS (Modified Ashworth Scale) and by patients using a VAS (Visual Analogue Scale)
Mobility will be assessed using the TUG scale (Time Up and Go) | This will be assessed through study completion, an average of 3 months (at Visits 1, 2, 3, 4, 5 and 6)
  TUG (Time Up and Go)is a validated test in patients with stroke. The score is expressed as the time (in seconds) required to perform sequential motor tasks (standing up from the chair, walking to the line on the floor at a normal pace, turning, walking back to the chair at a normal pace and finally sitting down).
Mobility will be assessed using the FES-I (Falls Efficacy Scale-International scale) | Evaluation will occur before Visit 5 (Day 60) and after Visit 6 (Day 90) 4 weeks of using EXOPULSE Mollii suit (Phase 2)
  Subjective risk of fall will be assessed using the French version of the Falls Efficacy Scale-International scale (FES-I) ; a 14-item scale that assesses the perceived risk of falling.
Quality of life will be measured using the EQ-5D-5L (EuroQol 5 Dimensions 5 Levels Quality of Life Questionnaire) | Evaluation will occur before Visit 5 (Day 60) and after Visit 6 (Day 90) 4 weeks of using EXOPULSE Mollii suit (Phase 2)
  This variable will be measured using the EuroQol 5 dimensions quality of life questionnaire, a scale developed by EuroQoL group. This scale has good psychometric properties in stroke and seems to be the most used generic health status questionnaire in this population. The 5 levels version (EQ-5D-5L) will be adopted in this work. The scale evaluates five dimensions: anxiety/depression, mobility, pain/difficulty, self-care, and usual activities.
Pain and fatigue will be assessed using a VAS (Visual Analogue Scale) | This will be assessed through study completion, an average of 3 months (at Visit 1, V2, V3, V4, V5 and V6)
  The visual analog scale for pain is a 10 mm straight line with one end meaning no pain and the other end meaning the worst pain imaginable
Evaluation of overall improvement using the CGI (Clinical Global Impression) | This will be assessed at Visit2 (Day 15) , Visit4 (Day 45) and Visit6 (Day 90) since CGI is designed to be applied after interventions
  It consists of 7-point scale ranging from "very much improved since the initiation of treatment" to "very much worse since the initiation of treatment" (from 1 to 7)
Evaluation of patient's blinding to the type of stimulation in the crossover trial | This will only be assessed at Visit2 (Day 15) and Visit4 (Day 45) since it's designed to be applied after interventions of phase 1 (double blind phase)
  This blind evaluation will be done in phase 1 using a dedicated questionnaire (only at visits 2 and 4 after each condition, as all patients will receive the same active treatment during open-label phase 2).

CONTACTS AND LOCATIONS:
Overall Officials: Samar S AYACHE, MD, PhD, Principal Investigator — Clinical Neurophysiology department, Henri Mondor Hospital, Creteil, France
Locations (1):
- Clinical Neurophysiology department, Henri Mondor Hospital, Creteil, France, Créteil, VAL DE MARNE, France